CLINICAL TRIAL: NCT01137903
Title: Prospective Randomized Clinical Trial Comparing Efficacy Surgical Versus Medical Treatment of Osteomyelitis in Diabetic Foot Ulcers
Brief Title: Efficacy of Surgical Treatment of Osteomyelitis in Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: José Luis Lázaro Martínez/Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OM-2010
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-05

CONDITIONS: Osteomyelitis; Diabetic Foot; Diabetic Foot Ulcers
Keywords: Diabetic foot; Osteomyelitis; Diabetic foot ulcers; Foot infections
MeSH Terms: conditions — Osteomyelitis; Diabetic Foot | interventions — Ciprofloxacin; Amoxicillin-Potassium Clavulanate Combination; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients undergoing medical treatment (Other): Antibiotic treatment within 90 days with:
  Ciprofloxacin Amoxicillin /Clavulanic acid. Trimethoprim /Sulfamethoxazole.
  Interventions: Drug: Ciprofloxacin; Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Sulfamethoxazole trimethoprim
- Patients undergoing surgical treatment (Other): Conservative surgical Minor amputation 7 days antibiotic after surgical
  Interventions: Procedure: Conservative surgery

INTERVENTIONS:
Procedure: Conservative surgery — Osteotomy, phalangectomy, exostectomy, metatarsal head resection, articular resection, partial calcanectomy
  Arms: Patients undergoing surgical treatment
Drug: Ciprofloxacin — 500 mg/ 12 hours during 90 days
  Arms: Patients undergoing medical treatment
Drug: Amoxicillin-Potassium Clavulanate Combination — 875/125 mg/12 hours during 90 days
  Arms: Patients undergoing medical treatment
Drug: Sulfamethoxazole trimethoprim — Trimethoprim 160 mg / Sulfamethoxazole 800 mg 1/12 horas.
  Arms: Patients undergoing medical treatment

SUMMARY:
Hypothesis:Surgical treatment of osteomyelitis in diabetic foot is more effective that medical treatment through antibiotherapy and leads wound healing in ulcers complicated with bone infection.Material and Methods: Randomized clinical trials which include two groups of patients (n=88), one receives medical treatment through antibiotherapy during 90 days and the other group receive conservative surgical treatment and antibiotics during 7 days after surgery. It will be studied differences between both groups in healing time, recidives, present and relationship of adverse events and outflow of quality of life related health .

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus Type 1 or 2.
* Patients with diabetic foot ulcers.
* Patients with clinical suspects of osteomyelitis.
* Patients with positive probe to bone test.
* Patients with signs of osteolysis in the bone located adjacent to the ulcer in X-Ray
* Patients with transcutaneous oxygen oxygenation above 30 mmHg.
* Acceptance to participate in the study through prior informed consent.

Exclusion Criteria:

* Patients with osteomyelitis associated with necrotizing soft tissue infections.
* Presence of necrotic tissue in the wound bed, edges or margins of the lesion.
* HbAc1 > 10.
* Presence of systemic toxicity such as fever, tachycardia, confusion, disorientation, vomiting or other signs usually related to systemic infection.
* Patients with bone exposure through the ulcer.
* Patients with absent pulses, ankle/brachial index (ABI) <0.8 and TcPO2 <30 mmHg.
* Pregnancy.
* Allergies to antibiotics.
* Any degree of renal impairment that contraindicated the administration of antibiotics proposed.
* Hepatic insufficiency.
* Mental Illnesses that prevent the understanding by the patient's proposed treatment, or for any other reason associated with your mental health, to recommend their inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Number of healing patients | 12 weeks
  Number of diabetic foot ulcers healing in both arms.

SECONDARY OUTCOMES:
Reulceration | 1 year after healing
  Analysis of re-ulceration events in both arms after healing in a 1 year follow-up
Healing time | 12 weeks
  Healing time in both arms
Complications | 12 weeks
  Percentage of complications in both arms
Quality of life | 12 weeks
  Quality of life related to health in both arms

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Lázaro Martínez, PhD, Principal Investigator — Universidad Complutense de Madrid; Francisco Javier Aragón Sánchez, MD, PhD, Study Chair — Hospital La Paloma Las Palmas de Gran Canaria
Locations (1):
- José Luis Lázaro Martínez, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lazaro-Martinez JL, Aragon-Sanchez J, Garcia-Morales E. Antibiotics versus conservative surgery for treating diabetic foot osteomyelitis: a randomized comparative trial. Diabetes Care. 2014;37(3):789-95. doi: 10.2337/dc13-1526. Epub 2013 Oct 15. PMID 24130347